CLINICAL TRIAL: NCT00426140
Title: An Open-label Single Center Study to Characterize the Absorption, Distribution, Metabolism, and Elimination (ADME) of Patupilone (EPO906) After a Single Intravenous Administration of 10 mg/m2 [14C] Patupilone in Patients With Advanced Solid Tumor Malignancies.
Brief Title: Pharmacokinetics of Patupilone After a Single Intravenous Administration in Patients With Advance Solid Tumor Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2122
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2010-04

CONDITIONS: Advanced Malignancies; Solid Tumors
Keywords: EPO; Patupilone; Solid Tumors
MeSH Terms: interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
The main purpose of this study is to characterize the distribution, metabolism, and elimination (ADME) of Patupilone after a single intravenous administration in patients with advanced solid tumor malignancies

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. World Health Organization (WHO) Performance Status Score of: 0- you are fully active and more or less as you were before your illness, 1 - you cannot carry out heavy physical work, but can do anything else.
3. Adequate hematological laboratory parameters
4. No major impairment of renal or hepatic function
5. Female patients must have a negative serum pregnancy test at screening.

Exclusion Criteria:

1. Severe and/or uncontrolled medical disease;
2. Severe cardiac insufficiency with uncontrolled and/or unstable cardiac or coronary artery disease;
3. Known diagnosis of human immunodeficiency virus (HIV) infection;
4. Presence of any other active or suspected acute or chronic uncontrolled infection;
5. Symptomatic brain metastases or leptomeningeal disease.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetic profile of patupilone including any potential metabolite(s) in blood/plasma as well as the total radioactivity in blood and plasma. | one week

SECONDARY OUTCOMES:
Safety and tolerability will be assessed by AEs, SAEs and out of range lab values. | every 6 weeks
Radiological scans will also be completed at approximately 6 weeks to asses anti-tumor activity. | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Cancer Therapy and Research Center, Institution for Drug Development, San Antonio, Texas, United States

REFERENCES:
- See also: Results can be found for CEPO906A2122 on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2941